CLINICAL TRIAL: NCT06562036
Title: Efficacy of Milrinone Plus Sildenafil in the Treatment of Neonates With Persistent Pulmonary Hypertension: A Single-Center, Randomized Controlled Trial
Brief Title: Efficacy of Milrinone With Sildenafil in Persistent Pulmonary Hypertension in Children
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Muhammad Aamir Latif (Other)
Responsible Party: Sponsor-Investigator, Muhammad Aamir Latif, Research Consultant, RESnTEC, Institute of Research
Organization: RESnTEC, Institute of Research (Other)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: DRAWAIS
Record Dates: First submitted 2024-08-17; First posted 2024-08-20 (Actual); Last update posted 2024-08-26 (Actual); Status verified 2024-08

CONDITIONS: Persistent Pulmonary Hypertension of the Newborn
MeSH Terms: conditions — Persistent Fetal Circulation Syndrome | interventions — Sildenafil Citrate; Milrinone

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Sildenafil (Experimental): Patients were given oral sildenafil at 2 mg per kg per day, 6-hourly, with an increment of 0.5 mg per kg per dose and a target maintenance dose of 2 mg per kg per dose every 6 hours by nasogastric tube.
  Interventions: Drug: Sildenafil
- Sildenafil + Milrinone (Experimental): In this group, Milrinone was initiated at 0.5 ug per kg per minute using intravenous infusion through a syringe pump, and sildenafil was given in the same protocol mentioned for the Sildenafil Group.
  Interventions: Drug: Sildenafil; Drug: Milrinone

INTERVENTIONS:
Drug: Sildenafil — Patients were given oral sildenafil as 2 mg per kg per day, 6-hourly with an increment of 0.5 mg per kg per dose and a target maintenance dose of 2 mg per kg per dose every 6 hour by nasogastric tube.
Drug: Milrinone — In this group, Milrinone was initiated at 0.5 ug per kg per minute using intravenous infusion through a syringe pump, and sildenafil was given in the same protocol mentioned for the Sildenafil Group.
  Arms: Sildenafil + Milrinone

SUMMARY:
Neonates with persistent pulmonary hypertension (PPH) should be administered inhaled nitric oxide (iNO) and extracorporeal membrane oxygenation (ECMO), but these are not available in most resource-constrained settings like ours. This study was planned to compare the outcomes of Milrinone plus Sildenafil versus Sildenafil alone in the treatment of PPH in neonates.

ELIGIBILITY:
Inclusion Criteria:

* Patients of either gender
* Aged between 1-28 days
* Birth weight above 2000 grams
* Diagnosed with persistent pulmonary hypertension (as per echocardiography)

Exclusion Criteria:

* Neonates having congenital heart defects (CHDs)
* Congenital diaphragmatic hernia
* Lung anomalies
* History of any surgical intervention

Ages: 1 Day to 28 Days | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 42 (Actual)
Dates: Start 2023-12-01 (Actual); Primary Completion 2024-05-31 (Actual); Study Completion 2024-05-31 (Actual)

PRIMARY OUTCOMES:
Change in pulmonary artery systolic pressure | 72 hours
  Efficacy was labeled yes if there was adecrease in pulmonary artery systolic pressure (PASP)

CONTACTS AND LOCATIONS:
Overall Officials: Muhammad Awais, FCPS, Principal Investigator — Children's Hospital and institute of Child Health Multan, Punjab, Pakistan; Abdur Rehman, FCPS, Study Director — Children's Hospital and institute of Child Health Multan, Punjab, Pakistan
Locations (1):
- Children's Hospital and institute of Child Health, Multan, Punjab Province, Pakistan

IPD SHARING:
Plan to Share IPD: No
Data can be shared with other researchers on a reasonable request